CLINICAL TRIAL: NCT02762461
Title: Artificial Reproductive Techniques (ART) and Progression of Endometriosis Symptoms
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: MMF2016
Record Dates: First submitted 2016-04-28; First posted 2016-05-05 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Endometriosis
Keywords: Fertilization in Vitro; Sperm Injections, Intracytoplasmic; Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Exposed group: Women with peritoneal/ovarian endometriosis and DIE (rectovaginal and rectosigmoid endometriosis) undergoing ART (IVF or ICSI).
  Interventions: Procedure: IVF or ICSI
- Reference group 1: Women with infertility because of factors other than endometriosis, e.g. male factor, undergoing ART (IVF or ICSI).
  Interventions: Procedure: IVF or ICSI
- Reference group 2: Women with medically treated endometriosis not undergoing ART.

INTERVENTIONS:
Procedure: IVF or ICSI
  Groups: Exposed group; Reference group 1

SUMMARY:
This project will investigate worsening of symptoms in endometriosis patients undergoing artificial reproductive techniques (ART). The study compares patients with peritoneal/ovarian and deep infiltrating endometriosis to relevant reference groups. Symptoms are monitored with a questionnaire with the categories quality of life, pain and bowel habits. The EHP-30® questionnaire is included in the questionnaire.

DETAILED DESCRIPTION:
Endometriosis affects up to 10% of all fertile women, and is associated with symptoms like infertility, dysmenorrhea, deep dyspareunia and chronic pelvic pain. 10-25% of endometriosis patients need artificial reproductive techniques (ART) to become pregnant. Endometriosis is estrogen dependent, and in theory this means, that the increased levels of estrogen during fertility treatment will worsen endometriosis symptoms. Endometriosis is a benign disease, and treatment is guided by the patient's symptoms. Worsening of endometriosis symptoms during fertility treatment may result in cessation of the treatment, operation and risk of complications.

This project will investigate worsening of symptoms in endometriosis patients undergoing artificial reproductive techniques (ART). The study compares endometriosis patients undergoing ART to two relevant reference groups; one group consisting women undergoing ART with infertility because of factors other than endometriosis, and one group consisting women with medically treated endometriosis not undergoing ART. Symptoms of endometriosis during ART will be monitored using a questionnaire that among other questions includes the validated questionnaire Endometriosis Health Profile 30® (EHP-30®). The questionnaire is administered before starting ART and later in the cycle before the patient gets to know if she is pregnant. The questionnaires as well as data collection will be administered electronically in REDCap® which is a secure web application for building and managing online surveys and databases.

ELIGIBILITY:
Inclusion Criteria:

* Female
* < 40 years
* Either undergoing ART (IVF or ICSI) with or without endometriosis or medically treated endometriosis

Exclusion Criteria:

* > 40 years

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Women with endometriosis under the age of 40 years.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Endometriosis Health Profile 30® (EHP-30®) | Groups undergoing ART: Change from baseline measures before stimulation during ART to ten days after aspiration. Reference group not undergoing ART: Change from baseline measures to four weeks later.
  The core instruments have five scale scores covering: Pain (11 questions), control and powerlessness (6 questions), social support (4 questions), emotional well-being (6 questions), self-image (3 questions).

SECONDARY OUTCOMES:
Pain (NRS scale: 0-10) | Groups undergoing ART: Change from baseline measures before stimulation during ART to ten days after aspiration. Reference group not undergoing ART: Change from baseline measures to four weeks later.
  Three categories with frequency, general, and worst perception of pain. In each category the patient has to rate her pain on the NRS scale according to dysmenorrhea, chronic pelvic pain, dyspareunia, defecation and urination pain. In addition there are qualitative questions in the same categories of pain.
Bowel habits | Groups undergoing ART: Change from baseline measures before stimulation during ART to ten days after aspiration. Reference group not undergoing ART: Change from baseline measures to four weeks later.
  Defecation frequency and time, stool consistency and blood in stool. Frequency and general perception of five bowel symptoms (constipation, diarrhea, nauseousness, emesis, and bloatedness) on a scale from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Mie Mathiasen, Student, Principal Investigator — University of Aarhus
Locations (1):
- Department of Gynaecology and Obstetrics, Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No